CLINICAL TRIAL: NCT05924451
Title: Study of Hard and Soft Tissue Behavior Around Abutments on Implants: Randomized Clinical Trial.
Brief Title: Study of Hard and Soft Tissue Behavior Around Abutments on Implants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Luis Carlos Garza Garza, Professor of Restorative Dentistry, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REST-ECL-2020-02
Record Dates: First submitted 2023-05-07; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous | interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned into two main groups according to the time of implant loading, in group A, an early loading will be applied with a PMMA and in group B, an immediate functional loading protocol will be applied with the zirconia prosthesis over the implants.
Who Masked: Investigator
Masking Description: The clinician performs the treatment of implant placement and prosthesis and the investigator analyzes the hard and soft tissue changes recorded over time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early loading (Active Comparator): The implants will be restored with a PMMA (polymethyl methacrylate) prosthesis in normal occlusion.
  Interventions: Behavioral: Immediate Loading
- Immediate loading (Experimental): The implants will be restored with a permanent prosthesis (monolithic zirconia) placed on the implants as an immediate loading.
  Interventions: Behavioral: Immediate Loading

INTERVENTIONS:
Behavioral: Immediate Loading — Clinical and radiographic examination of the periimplant soft and hard tissue will be analysed by using gingival index, plaque index, and pocket depth immediately post operative.

SUMMARY:
Purpose: To compare the loss of peri-implant tissue by means of radiographic and digital analysis of a zirconia prosthesis placed immediately and delay loading.

Materials and methods: 60 consecutive patients with the need for a full-arch rehabilitation were selected and divided randomly into two groups:

Group A: Conventional dental extraction, placement of 6 to 8 implants. Placement of the multi-unit prosthetic attachment and finally in the same week the placement of the definitive monolithic zirconia prosthesis on implants. Group B: Conventional dental extraction, placement of 6 to 8 implants. Placement of prosthetic and provisional attachment. After 3 months, place the definitive prosthesis. Assess volumetric changes using radiographic and optical scan techniques.

The number of implant failures, prosthetic incidents and bone loss around the implants will be evaluated. The data will be evaluated 3, 6, and 12 months after the operation.

DETAILED DESCRIPTION:
All patients volunteered will be selected from the Clinica Universitaria de Odontología (CUO) of the Universitat Internacional de Catalunya (Spain) and also from the Clinica Dental Crooke & Laguna to participate in the study must sign an informed consent form based on the Helsinki Declaration of 1975, as revised in 2013. The patients must required implants for implant-supported restorations and will be thoroughly informed regarding the nature of the study. This study will include 60 patients. The sample number required for the study was determined with an alpha risk of 0.05, a power of 80%, a standard deviation of 1.1mm and estimating a loss rate to follow-up of 20%.

In this prospective cohort multi-centric clinical study all implants of the same brand will be tested. The study will be conducted in the Clinica Universitaria de Odontologia from the Universitat Internacional de Catalunya located in C/ Josep Trueta, s/n, 08195 Sant Cugat del Vallès and also in the Clinica Dental Crooke Marbella located in Calle Mediterráneo, 1. 29602 Marbella (Málaga)

On the surgical and prosthetic protocols will be performed by experienced clinicians in accordance to the manufacturer's recommendations. All surgical procedures will be conducted under local anesthesia (Ultracain; Aventis Inc., Frankfurt, Germany). Sinus augmentation procedures will be performed in patients with inadequate bone availability, applying the bone scraper technique as described elsewhere. All sinus cavities will be grafted using autologous cortical bone in combination (approximate ratio of 1:1) with anorganic bovine bone particles (250-1000 lm in size, Bio-Oss; Geistlich Pharma AG, Wolhusen, Switzerland) and a healing period of six to nine months is required for implant placement.

A conventional implant placement protocol using only Nobel Parallel Implants will be followed in patients not requiring maxillary sinus augmentation. The maxilla or mandible will be surgically exposed. Any resining compromise teeth will be removed either before or after flap elevation based on the surgeon's preference. The bony platform of the residual mandible will be surgically levelled parallel to the opposing occlusal plane to create a space for the restoration and/or soft tissue. Analog drill guides and templates will be used to ensure precise placement of implants in the correct location while accommodating the position of the dentition.

All patients will be prescribed a pharmacologic regimen of amoxicillin/clavulanic acid tablets (875/125 mg, TID for 7 days) or, if allergic to penicillin, clindamycin tablets (300 mg, TID for 7 days), and anti-inflammatory medication (Ibuprofen 600 mg every 4 to 6 hours as needed to a maximum of 3600 mg/ day). Six implant pure titanium (grade IV) dental implants with an acid-etched surface will be used.

Patients will be divided into two main groups according to the time of implant loading:

1. Group A (n=30) - An early loading will be applied. Implants receive early loading protocol where temporary framework with a PMMA (poly-methyl methacrylate) will be fabricated in normal occlusion.
2. Group B (n=30) - An immediate functional loading protocol will be applied. A permanent framework (monolithic Zirconia) will be placed in mouth over implants.

Clinical examination of the implant soft tissue will be done using gingival index, plaque index, and pocket depth immediately post operative, at 3, 6 and 12 months after the operation.

Standardized digital periapical radiographs (Kodak ACR-2000; Eastman Kodak Company, Rochester, NY, USA) will be obtained at the time of treatment planning, after implant surgery (baseline), at 1, 3, 6 and 12 months intervals. They will be exported to a computer software package for further analysis (Dent-A-View v1.0; DigiDent, DIT, Nesher, Israel). For the MBL determination, a single independent calibrated examiner will made linear measurements on each periapical radiograph from the most mesial and distal point of the implant platform to the crestal bone. The magnification of the radiograph will be corrected in accordance with the clinical data (height and width) for each implant. To calibrate each linear marginal bone loss a simple mathematical calculation will be performed and measured according to the radiographic image size.

Data will be gathered of all patients on a database so the identity of the patient is not compromised, the information collected will contain their age, gender, tobacco and alcohol consumption habits (at the time of study enrollment), history of periodontal disease, and bone substratum. Smoking status will be classified as non-smoker (0 cig/day), mild smoker (0-10 cig/day), and heavy smoker (>10 cigs/day). Patients with an alcohol intake >10 g/day will be considered alcohol consumers. Periodontal disease history will be determined by assessment of the clinical attachment loss (CAL) using a Michigan O probe (Hu-Friedy, Chicago, IL, USA): patients with ≥4 sites exhibiting CAL ≥3 mm (excluding third molars) will be considered to have periodontitis.

After a descriptive statistical analysis, a linear mixed model will be used to determine the effects of abutment height and platform switching on the MBL at two peri-implant sites (mesial and distal) at 1, 3, 6 and 12 months intervals after transmucosal abutment placement, controlling for age, gender, smoking habits, periodontal status, prosthesis type, bone substratum type, and implant length. A scaled identity covariance matrix will be used, following Schwarz Bayesian information criterion. Significant difference will be found between mesial and distal aspects or between time points, the average MBL values will be used to reveal the effects of the variables of interest.

The Gingival Index will be assessed according to a modified version of Loe and Silness and scored as: 0 = normal mucosa, 1 = bleeding with superficial probing, or 2 = spontaneous bleeding. The bleeding tendency will be assessed using a modified Sulcus Bleeding Index (mBI) according to Mombelli et al. and scored as: 0 = no bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant, 1 = isolated bleeding spots visible, 2 = blood forms a confluent red line on the margin, or 3 = heavy or profuse bleeding. The status of the keratinized mucosa surrounding the implant will be evaluated as: 0 = no keratinized mucosa around the implant, 1 = mucosa surrounding the implant is partially keratinized, or 2 = the entire mucosa surrounding the implant is keratinized.

Patient satisfaction will be evaluated separately in function and esthetics using a scale with ratings of 0 to 10 where 10 = fully satisfied and 0 = not satisfied. The clinicians' assessment will be based on their impression of the treatment concept. The clinician scored function and esthetics separately from 1 to 10, with 10 = excellent, 5 = average, and 1 = poor.

Descriptive statistics, including frequency tables, mean values, and standard deviations, will be used to present the results. Statistical analyses will be performed using SPSS Statistics Desktop software version 24.0 (SPSS).

ELIGIBILITY:
Inclusion Criteria of the subjects:

* At least 18 years of age
* Physically and mentally capable of completing the 1-year follow-up
* With a stable occlusal relationship with or without opposing dentition
* Are willing and able to comply with study-related procedures
* Have good oral hygiene
* Present good quality and quantity of bone for implant placement.
* Must be American Society of Anesthesiologists (ASA) physical status of I or II, periodontal stable, and can enroll in a periodontal maintenance program.

Exclusion Criteria:

* Health conditions that do not permit surgical or restorative procedures (including anesthesia).
* Disorder in the planned implant area (eg, previous tumors, chronic bone disease, or previous irradiation).
* History of alcohol or drug abuse
* Smoke more than one pack of cigarettes per day (> 20 cigarettes or equivalent)
* Uncontrolled diabetes
* Bisphosphonate therapy
* Pathologic occlusion, (eg, severe bruxism or other parafunctional habits)
* Lack opposing dentition or has unstable occlusion
* Needs of bone augmentations or sinus lift treatments
* Ongoing infections or endodontic or periodontal problems in opposing teeth or implants
* Poor oral hygiene
* Allergic or adverse reactions to the restorative material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Overall result of final prosthesis | One day
  The final prosthesis will be judged by the patient. A 10 cm Visual analogue scale (VAS) is used. 0 (unacceptable) is placed in left end, and 10 (perfect) is placed in the right end.
Gingival index | One day
  The Gingival Index will be assessed according to a modified version of Loe and Silness and scored as: 0 = normal mucosa, 1 = bleeding with superficial probing, or 2 = spontaneous bleeding.
Patient satisfaction | One day
  Patient satisfaction will be evaluated separately in function and esthetics using a scale with ratings of 0 to 10 where 10 = fully satisfied and 0 = not satisfied.
Bone-implant contact | One day
  A single independent calibrated examiner will made linear measurements on each periapical radiograph from the most mesial and distal point of the implant platform to the crestal bone.

CONTACTS AND LOCATIONS:
Overall Officials: MIGUEL ROIG CAYON, MD DDS PHD, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Clinica Universitaria d'Odontologia, Sant Cugat Del Vallés, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
All data will be published

REFERENCES:
- [Background] Gomez-Polo M, Ballesteros J, Perales-Padilla P, Perales-Pulido P, Gomez-Polo C, Ortega R. Guided implant scanning: A procedure for improving the accuracy of implant-supported complete-arch fixed dental prostheses. J Prosthet Dent. 2020 Aug;124(2):135-139. doi: 10.1016/j.prosdent.2019.09.022. Epub 2019 Nov 21. PMID 31761274
- [Background] Suarez-Feito JM, Sicilia A, Angulo J, Banerji S, Cuesta I, Millar B. Clinical performance of provisional screw-retained metal-free acrylic restorations in an immediate loading implant protocol: a 242 consecutive patients' report. Clin Oral Implants Res. 2010 Dec;21(12):1360-9. doi: 10.1111/j.1600-0501.2010.01956.x. PMID 20637035
- [Background] Meneghetti P, Moura GF, Tavelli L, Li J, Siqueira R, Wang HL, Mendonca G. A fully digital approach for implant fixed complete dentures: A case report. J Esthet Restor Dent. 2021 Dec;33(8):1070-1076. doi: 10.1111/jerd.12798. Epub 2021 Jul 2. PMID 34213055
- [Background] Espona J, Roig E, Ali A, Roig M. Immediately loaded interim complete-arch implant-supported fixed dental prostheses fabricated with a completely digital workflow: A clinical technique. J Prosthet Dent. 2020 Oct;124(4):423-427. doi: 10.1016/j.prosdent.2019.08.008. Epub 2019 Dec 18. PMID 31862143